CLINICAL TRIAL: NCT02183909
Title: Connecting Resources for Urban Sexual Health
Acronym: CRUSH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EI12-EBACA-003
Record Dates: First submitted 2014-05-06; First posted 2014-07-08 (Estimated); Results first posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: HIV; Sexually Transmitted Infections
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study intervention (Experimental)
  Interventions: Other: Testing and linkage to care for Y/MSM; Behavioral: Engagement and retention for HIV-positive Y/MSM in care; Other: Engagement and retention for HIV-negative Y/MSM in sexual health services; Drug: Stribild PEP Substudy

INTERVENTIONS:
Other: Testing and linkage to care for Y/MSM — Implementation of strategies to enhance testing and linkage to care of Y/MSM, including social network testing and a youth outreach corps working with existing and new community partner agencies.
Behavioral: Engagement and retention for HIV-positive Y/MSM in care — Optimizing current HIV care and treatment services at DYC by implementing a patient peer mentoring component, a linkage and retention specialist, and psychosocial support for program staff.
Other: Engagement and retention for HIV-negative Y/MSM in sexual health services — Offering a highly effective combination HIV prevention strategy, including PrEP; warm-hand offs for high-risk negatives, nPEP; risk reduction counseling; frequent HIV and STI testing, including testing a highly sensitive method of detecting early HIV infection; and youth-focused programming.
Drug: Stribild PEP Substudy — A substudy of 28 days of once-daily Stribild® initiated within 72 hours of a high risk sexual exposure for HIV post-exposure prophylaxis (PEP).

SUMMARY:
The overall goal of the CRUSH project is to enhance and extend a response to the local HIV/AIDS epidemic in Alameda County with a set of innovative, evidence-based interventions across the continuum of HIV prevention and care, targeting individuals and communities most vulnerable to HIV. The East Bay AIDS Center, in partnership with the University of California San Francisco's Center for AIDS Prevention Studies, the Gladstone Institutes, and several key community-based organizations, are engaging in a participatory partnership to enhance and implement HIV services which target the East Bay's highest risk population- young men who have sex with men (Y/MSM). Specifically, the CRUSH Project is designed to evaluate a combination of program approaches to address the sexual health care needs of young gay men of color and their sexual partners by enhancing the current program activities of the Downtown Youth Clinic (DYC).

We hypothesize that we can reduce the impact of HIV among Y/MSM by expanding the current DYC services structure in two ways. We intend to expand HIV testing, and linkage to and retention in care for youth who test HIV positive, providing them with intensive risk-reduction counseling and antiretroviral treatment, and thereby ultimately reducing the risk of further HIV transmission. And we intend for the first time to offer a comprehensive combination package of preventive services to HIV-negative youth, including routine accesses to HIV/STI screening and treatment, and access to HIV pre-exposure prophylaxis (PrEP).

The CRUSH Project will also have a substudy that will enroll HIV-negative participants who are eligible to receive PEP. The substudy will evaluate the tolerability and acceptability of a 28 day course of Stribild® given as post-exposure prophylaxis (PEP) to prevent sexual acquisition of HIV-1 in Y/MSM of color.

DETAILED DESCRIPTION:
The CRUSH Project (Connecting Resources for Urban Sexual Health) is a demonstration project at Alta Bates Summit Medical Center's East Bay AIDS Center (EBAC) and Downtown Youth Clinic (DYC) offering interventions aimed at reducing HIV-1 incidence among young MSM of color in the East Bay region. CRUSH has two major components:

1. Providing enhanced testing and linkage to care (TLC+) for HIV positives, aimed at increasing the proportion of HIV positive Y/MSM who are in care, virologically suppressed, and receiving intensive risk reduction counseling.
2. Providing comprehensive sexual health services to high risk HIV-negatives, including but not limited to the provision of PrEP and PEP when clinically appropriate.

In addition, the CRUSH Project will offer a substudy of CRUSH, and will enroll HIV negative CRUSH participants who are eligible to receive PEP. Stribild® is a single-tablet, four-drug, once-daily complete regimen that is FDA-approved for the treatment of HIV-1 infection in treatment-naïve HIV-infected adults with estimated glomerular filtration rate ≥70ml/min/1.73m2. Because of limited data, no antiretroviral drug or combination of drugs has been approved for PEP. Current PEP guidelines generally call for using a 28-day course of a 3-drug regimen that has been approved for the treatment of HIV-1 infection

ELIGIBILITY:
Inclusion Criteria:

* Men between the ages of 18-29 who are ever sexually active with men;
* Transgender females (M2F) between the ages of 18-29 who are sexually active with men; Transgender males (F2M) between the ages of 18-29 who are sexually active with men; and
* Any HIV-negative person aged 18-29, male or female, who has at least one known HIV positive (i.e. serodiscordant) sexual partner.

Exclusion Criteria:

* None.

For the PEP substudy the inclusion criterion is at least one episode in the 72 hours prior to presentation of unprotected receptive anal intercourse with a partner known or suspected to be HIV positive and the following are the substudy exclusion criteria:

* Known kidney disease
* Dipstick proteinuria >1+
* eGFR < 70 ml/min/1.73m2
* Known metabolic bone disease
* Signs or symptoms of acute HIV infection
* Concomitant use of nephrotoxic drug or medication contraindicated with Stribild®

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 378 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Burack, MD, Principal Investigator — East Bay AIDS Center (EBAC); Robert Grant, MD, MPH, Principal Investigator — Gladstone Institutes; Janet Myers, PhD, Principal Investigator — UCSF Center for AIDS Prevention
Locations (1):
- Downtown Youth Clinic, Oakland, California, United States

REFERENCES:
- [Background] Grant RM, Lama JR, Anderson PL, McMahan V, Liu AY, Vargas L, Goicochea P, Casapia M, Guanira-Carranza JV, Ramirez-Cardich ME, Montoya-Herrera O, Fernandez T, Veloso VG, Buchbinder SP, Chariyalertsak S, Schechter M, Bekker LG, Mayer KH, Kallas EG, Amico KR, Mulligan K, Bushman LR, Hance RJ, Ganoza C, Defechereux P, Postle B, Wang F, McConnell JJ, Zheng JH, Lee J, Rooney JF, Jaffe HS, Martinez AI, Burns DN, Glidden DV; iPrEx Study Team. Preexposure chemoprophylaxis for HIV prevention in men who have sex with men. N Engl J Med. 2010 Dec 30;363(27):2587-99. doi: 10.1056/NEJMoa1011205. Epub 2010 Nov 23. PMID 21091279
- [Background] Baeten JM, Donnell D, Ndase P, Mugo NR, Campbell JD, Wangisi J, Tappero JW, Bukusi EA, Cohen CR, Katabira E, Ronald A, Tumwesigye E, Were E, Fife KH, Kiarie J, Farquhar C, John-Stewart G, Kakia A, Odoyo J, Mucunguzi A, Nakku-Joloba E, Twesigye R, Ngure K, Apaka C, Tamooh H, Gabona F, Mujugira A, Panteleeff D, Thomas KK, Kidoguchi L, Krows M, Revall J, Morrison S, Haugen H, Emmanuel-Ogier M, Ondrejcek L, Coombs RW, Frenkel L, Hendrix C, Bumpus NN, Bangsberg D, Haberer JE, Stevens WS, Lingappa JR, Celum C; Partners PrEP Study Team. Antiretroviral prophylaxis for HIV prevention in heterosexual men and women. N Engl J Med. 2012 Aug 2;367(5):399-410. doi: 10.1056/NEJMoa1108524. Epub 2012 Jul 11. PMID 22784037
- [Background] Thigpen MC, Kebaabetswe PM, Paxton LA, Smith DK, Rose CE, Segolodi TM, Henderson FL, Pathak SR, Soud FA, Chillag KL, Mutanhaurwa R, Chirwa LI, Kasonde M, Abebe D, Buliva E, Gvetadze RJ, Johnson S, Sukalac T, Thomas VT, Hart C, Johnson JA, Malotte CK, Hendrix CW, Brooks JT; TDF2 Study Group. Antiretroviral preexposure prophylaxis for heterosexual HIV transmission in Botswana. N Engl J Med. 2012 Aug 2;367(5):423-34. doi: 10.1056/NEJMoa1110711. Epub 2012 Jul 11. PMID 22784038

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Intervention: Testing and linkage to care for YMSM: Implementation of strategies to enhance testing and linkage to care of YMSM, including social network testing and a youth outreach corps working with existing and new community partner agencies. Engagement and retention for HIV-positive YMSM in care: Optimizing current HIV care and treatment services at DYC by implementing a patient peer mentoring component, a linkage and retention specialist, and psychosocial support for program staff. Engagement and retention for HIV-negative YMSM in sexual health services: Offering a highly effective combination HIV prevention strategy, including PrEP; warm-hand offs for high-risk negatives, nPEP; risk reduction counseling; frequent HIV and STI testing, including testing a highly sensitive method of detecting early HIV infection; and youth-focused programming. Stribild PEP Substudy: 28 days of once-daily Stribild® initiated within 72 hours of a high risk sexual exposure for HIV post-exposure prophylaxis (PEP).
Period: Overall Study
Arm/Group | Study Intervention
Started | 378 (378 were assessed for enrollment)
Completed | 324
Not Completed | 54

BASELINE CHARACTERISTICS:
Population: There were 98 HIV positive individuals and 23 HIV- individuals who were female or transgender who were excluded from the primary analyses of HIV negative YMSM.
Groups:
- HIV Negative YMSM: Testing and linkage to care for YMSM: Implementation of strategies to enhance testing and linkage to care of YMSM, including social network testing and a youth outreach corps working with existing and new community partner agencies. Engagement and retention for HIV-negative YMSM in sexual health services: Offering a highly effective combination HIV prevention strategy, including PrEP; warm-hand offs for high-risk negatives, nPEP; risk reduction counseling; frequent HIV and STI testing, including testing a highly sensitive method of detecting early HIV infection; and youth-focused programming. Stribild PEP Substudy: 28 days of once-daily Stribild® initiated within 72 hours of a high risk sexual exposure for HIV post-exposure prophylaxis (PEP).
Arm/Group | HIV Negative YMSM
Number analyzed (Participants) | 257
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.2 (2.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 257
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 40
  Latino | 84
  White | 64
  Asian | 33
  Other | 2
  Mixed | 17
  Refused/no response | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 257
Self-reported sexual orientation [Count of Participants; unit: Participants]
  Straight | 3
  Gay | 29
  Bisexual | 217
  Other | 7
  Refused to answer | 1
Highest level of education [Count of Participants; unit: Participants]
  High school or less | 65
  Some education post-high school | 188
  Missing | 4
Household is receiving public assistance [Count of Participants; unit: Participants]
  No Response/missing | 6
  No | 222
  Yes | 29
Health insurance in the past [Count of Participants; unit: Participants]
  None | 13
  Public Insurance | 38
  Private Insurance | 110
  Other Coverage | 69
  Multiple Types reported | 27
Received PEP at baseline visit [Count of Participants; unit: Participants]
  No | 227
  Yes | 30
Mental health (BSI screen symptomatic) [Count of Participants; unit: Participants]
  No | 254
  Yes | 2
  Missing data | 1
No. of sex partners Mean in past 3 mo [Mean (Standard Deviation); unit: Sex partners] | 7.65 (8.1)
No. of survival-related needs [Mean (Standard Deviation); unit: Number of competing needs reported] — Survival concerns were measured using questions adapted from the iPrEx-OLE study, and an index was created by adding the number of factors participants said affected their adherence.
  Number of competing needs reported | 0.55 (0.98)
Exposure to gun violence (ever) [Count of Participants; unit: Participants] | 38

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Young Men Who Have Sex With Men (YMSM) Who Test Positive for HIV at Enrollment
Description: Expanding the investigators currently successful HIV testing strategy-collaborations and systems of referral of new cases of HIV from existing partners-so that referrals are also received for high risk negatives to receive sexual health services. Implementing two new strategies: social network testing and a youth outreach corps working with partner agencies; it is hypothesized that social network testing will increase the proportion of positive test results.
Time Frame: 1 year
Population: The analysis population is all individuals who completed an enrollment process.
Measure: Count of Participants; unit: Participants
Groups:
- Study Intervention: Testing and linkage to care for Y/MSM: Implementation of strategies to enhance testing and linkage to care of Y/MSM, including social network testing and a youth outreach corps working with existing and new community partner agencies. Engagement and retention for HIV-positive Y/MSM in care: Optimizing current HIV care and treatment services at DYC by implementing a patient peer mentoring component, a linkage and retention specialist, and psychosocial support for program staff.
  Engagement and retention for HIV-negative Y/MSM in sexual health services: Offering a highly effective combination HIV prevention strategy, including PrEP; warm-hand offs for high-risk negatives, nPEP; risk reduction counseling; frequent HIV and STI testing, including testing a highly sensitive method of detecting early HIV infection; and youth-focused programming.
  Stribild PEP Substudy: A substudy of 28 days of once-daily Stribild® initiated within 72 hours of a high risk sexual exposure for HIV post-ex
Arm/Group | Study Intervention
Number analyzed (Participants) | 378
Participants
  Previously in care | 70
  Newly in care at CRUSH | 28
  HIV negative | 280

2. Primary Outcome: The Proportion of HIV-positive Enrolled YMSM Who Are Retained, on Therapy, and Who Have Achieved Viral Suppression Within One Year of Entering Care
Description: Optimizing current HIV care and treatment services at DYC by adding three new components: a patient peer mentoring component, a linkage and retention specialist, and psychosocial support for program staff.
Time Frame: 1 year
Population: HIV positive individuals in the CRUSH study.
Measure: Count of Participants; unit: Participants
Groups:
- HIV Infected Individuals: Engagement and retention for HIV-positive Y/MSM in care: Optimizing current HIV care and treatment services at DYC by implementing a patient peer mentoring component, a linkage and retention specialist, and psychosocial support for program staff.
Arm/Group | HIV Infected Individuals
Number analyzed (Participants) | 98
Participants
  Retained at 1 year | 81
  On Therapy at 1 year | 52
  Viral suppression | 47

3. Primary Outcome: The Proportion of HIV-uninfected YMSM Participants Who Are Retained, Receive Sexually Transmitted Infection (STI) Testing, and Receive Non-occupational Post-exposure-prophylaxis (nPEP) and/or PrEP
Description: Integrating sexual health services for HIV-uninfected young MSM of color into an HIV care setting, including PrEP, warm-hand offs for high risk negatives, nPEP, risk reduction counseling, frequent HIV and STI testing, and youth-focused programming.
Time Frame: 1 year
Population: All HIV negative YMSM who enrolled in the CRUSH study.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Negative YMSM
Number analyzed (Participants) | 257
Participants
  Retained: Yes | 243
  Retained: No | 14
  Received STI testing: Yes | 188
  Received STI testing: No | 69
  Received PrEP: Yes | 239
  Received PrEP: No | 18
  Received PEP: Yes | 30
  Received PEP: No | 227

4. Primary Outcome: Substudy Primary Outcome: The Tolerability and Acceptability of a 28 Day Course of Stribild® Given as Post-exposure Prophylaxis (PEP) to Prevent Sexual Acquisition of HIV-1
Description: Regimen completion at 28 days.
Time Frame: 4 Weeks
Population: 100 participants enrolled in the Stribild® sub study.
Measure: Count of Participants; unit: Participants
Groups:
- Stribild PEP Substudy: 28 days of once-daily Stribild® initiated within 72 hours of a high risk sexual exposure for HIV post-exposure prophylaxis (PEP).
Arm/Group | Stribild PEP Substudy
Number analyzed (Participants) | 100
Participants | 69

5. Secondary Outcome: Substudy Secondary Outcome: The Renal Safety of Stribild® PEP
Description: Change from week 1 to week 4 in serum creatinine.
Time Frame: 1 Week and 4 Weeks
Population: The number of participants with data available for this measure at four weeks.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Stribild PEP Substudy
Number analyzed (Participants) | 30
mg/dl | .0380 (.10855)

6. Secondary Outcome: Substudy Secondary Outcome: Change From 1 Week to 4 Weeks in eGFR
Description: To Assess the Renal Safety of Stribild® PEP. Change from 1 Week to 4 Weeks in estimated glomerular filtration rate (eGFR), which measures how well the kidneys are filtering waste and toxins from the blood.
Time Frame: 1 Week and 4 Weeks
Population: The number of participants with data available for this measure at four weeks.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m2
Arm/Group | Stribild PEP Substudy
Number analyzed (Participants) | 28
mL/min/1.73m2 | -1.4286 (10.86424)

7. Secondary Outcome: Substudy Secondary Outcome: To Assess the Renal Safety of Stribild® PEP
Description: Markers of proximal tubulopathy (glycosuria, proteinuria > 1+).
Time Frame: 4 Weeks
Population: 100 participants enrolled in the Stribild® sub study.
Measure: Count of Participants; unit: Participants
Arm/Group | Stribild PEP Substudy
Number analyzed (Participants) | 100
Participants | 0

8. Secondary Outcome: Substudy Secondary Outcome: To Document Any HIV-1 Seroconversions Occurring While on Stribild® PEP
Description: HIV-1 seroconversion.
Time Frame: 4 Weeks
Population: 23 participants did not return for the week 4 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Stribild PEP Substudy
Number analyzed (Participants) | 77
Participants | 0

9. Secondary Outcome: Substudy Secondary Outcome: To Assess Adherence to Stribild® PEP
Description: Self-reported adherence.
Time Frame: 4 Weeks
Population: 100 participants enrolled in the Stribild® sub study.
Measure: Count of Participants; unit: Participants
Arm/Group | Stribild PEP Substudy
Number analyzed (Participants) | 100
Participants | 69

10. Secondary Outcome: Substudy Secondary Outcome: To Assess Adherence to Stribild® PEP
Description: Reported reasons for non-adherence
Time Frame: 4 Weeks
Population: 69 substudy participants provided responses regarding reasons for adherence.
Measure: Count of Participants; unit: Participants
Arm/Group | Stribild PEP Substudy
Number analyzed (Participants) | 69
Participants
  Reasons for any non-adherence | 69
  Didn't have pills with me | 36
  Forgot to take my pills | 53
  Didn't feel like taking it | 2
  Schedule changes | 42
  Wanted to take it privately | 9
  Side-effects or feeling ill | 13
  Planned to drink/get high | 7
  I was drunk/high | 4
  Felt too emotional (sad, angry, anxious) | 7
  Was saving them for later | 1

11. Secondary Outcome: Substudy Secondary Outcome: To Assess Adherence to Stribild® PEP
Description: Changes from baseline in quality of life.
Time Frame: 4 Weeks
Population: Data were not collected for the quality of life measure.
Arm/Group | Stribild PEP Substudy
Number analyzed (Participants) | 0

12. Secondary Outcome: Substudy Secondary Outcome: To Assess Adherence to Stribild® PEP
Description: Early cessation of regimen.
Time Frame: 4 Weeks
Population: 100 participants enrolled in the Stribild® sub study.
Measure: Count of Participants; unit: Participants
Arm/Group | Stribild PEP Substudy
Number analyzed (Participants) | 100
Participants | 11

ADVERSE EVENTS:
Time Frame: up to 1 year for each participant
Arm/Group | Study Intervention
All-Cause Mortality (participants affected / at risk) | 0/378
Serious Adverse Events (participants affected / at risk) | 0/378
Other Adverse Events (participants affected / at risk) | 0/378

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2013-12-17): https://cdn.clinicaltrials.gov/large-docs/09/NCT02183909/Prot_000.pdf
  • Statistical Analysis Plan (2013-12-17): https://cdn.clinicaltrials.gov/large-docs/09/NCT02183909/SAP_001.pdf